CLINICAL TRIAL: NCT03776019
Title: Efficacy of Audio-Visual-Perception-Enhancement (AVWF®) Method in Chronic Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinikum Klagenfurt am Wörthersee (Other)
Responsible Party: Principal Investigator, Rudolf Likar, Prim.Univ.Prof.Dr., Klinikum Klagenfurt am Wörthersee
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AVWF 2019
Record Dates: First submitted 2018-12-10; First posted 2018-12-14 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Pain; Stress
Keywords: Pain; Stress; AVWF; Audio-Visual-Perception-Enhancement
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modulated (Experimental): modulated music
  Interventions: Device: AVWF device
- Typical (Sham Comparator): typical music
  Interventions: Device: AVWF device

INTERVENTIONS:
Device: AVWF device — The AVWF method utilizes sound modulated music, which is thought to regulate the vagus nerve.

SUMMARY:
It is anticipated that Audio-Visual-Perception-Enhancement (AVWF®) method leads to pain reduction and a decrease of inflammatory markers in chronic pain patients. Also an improvement of quality of life, self-perceived disability and depression in chronic pain patients is expected.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain with a numeric rating scale of pain >= 4 for > 6 month
* patients >18 years

Exclusion Criteria:

* psychosis
* drug addiction
* pension process
* pregnant women
* epilepsy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Numeric Rating Scale of Pain Severity | Change from baseline Numeric Rating Scale of Pain Severity after 10 interventions, 4 weeks after the last intervention, and 3 month after the last intervention
  Validated 11 pt scale 0-10, to evaluate a patient's current severity of pain. A rating of 0 indicates no pain while 10 indicates the worst pain imaginable. A score of 4 or above is considered a clinically significant pain Level.

SECONDARY OUTCOMES:
Health related quality of life | Change from baseline health related quality of life after 10 interventions, 4 weeks after the last intervention, and 3 month after the last intervention
  Health related quality of life will be measured by euroQol-5D questionnaire. It contains two sections, a descriptive section and a valuation section
Hospital Anxiety and Depression Scale | Change from baseline Hospital Anxiety and Depression Scale after 10 interventions, 4 weeks after the last intervention, and 3 month after the last intervention
  Anxiety and depression is evaluated by the the Hospital Anxiety and Depression Scale.It contains 14 items describing symptoms of depression (7 items) and anxiety (7 items). It was developed to identify anxiety and depression in non-psychiatric medical outpatients. Each item on the HADS is scored from 0 (no problem) to 3 (maximum distress).
Pittsburgh Sleep Quality Index | Change from baseline Pittsburgh Sleep Quality Index after 10 interventions, 4 weeks after the last intervention, and 3 month after the last intervention
  Self-report questionnaire that assesses sleep Quality through the measure of 19 individual items, creating 7 components that produce one global score
Depression Anxiety Stress Scales | Change from baseline Depression Anxiety Stress Scales after 10 interventions, 4 weeks after the last intervention, and 3 month after the last intervention
  A 42-item self report instrument designed to measure the three related negative emotional states of depression, anxiety and tension/stress.
Pain Disability Index | Change from baseline Pain Disability Index after 10 interventions, 4 weeks after the last intervention, and 3 month after the last intervention
  The Pain Disability Index is an instrument for measuring the impact that pain has on the ability of a person to participate in essential life activities. Minimal index: 0; maximal index: 70; The higher the index the greater the person's disability due to pain
Salival Cortisol level | Change from baseline salival cortisol level after 10 interventions, 4 weeks after the last intervention, and 3 month after the last intervention
  Immunoassay for in vitro quantitative determination of cortisol in saliva

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Likar, Principal Investigator — Head of department
Locations (1):
- Klinikum Klagenfurt am Wörthersee, Klagenfurt, Austria

IPD SHARING:
Plan to Share IPD: No